CLINICAL TRIAL: NCT07099118
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics of Single and Multiple Doses of HEC169584 Capsules and the Effect of Food on Its Pharmacokinetics in Healthy Subjects
Brief Title: A Safety, Tolerability, Pharmacokinetics/Pharmacodynamics Study of HEC169584 Capsules in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC169584-NASH-101
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Non - Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ascending Single and Multiple Dose Study is Double-blind design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Dose group-1 (Experimental): On day1 subjects will take the experiment drug on an empty stomach with 240ml warm water.
  Interventions: Drug: HEC169584 capsule
- Dose group-2 (Sham Comparator): Single ascending-dose study: on day1 subjects will take the 30 mg experiment drug on an empty stomach with 240ml warm water ;
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-3 (Sham Comparator): Single ascending-dose study: on day1, subjects will take 70 mg the experiment drug or placeble on an empty stomach with 240ml warm water.
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-4 (Sham Comparator): Single ascending-dose study: on day1, subjects will take 150 mg the experiment drug or placeble on an empty stomach with 240ml warm water.
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-5 (Sham Comparator): Single ascending-dose study: on day1, subjects will take 300 mg the experiment drug or placeble on an empty stomach with 240ml warm water. Subjects also need to take experiment drug after high - fat and high - calorie meals on day 15
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-6 (Sham Comparator): Single ascending-dose study: on day1, subjects will take 450 mg the experiment drug or placeble on an empty stomach with 240ml warm water.
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-7 (Sham Comparator): Single ascending-dose study: on day1, subjects will take 600 mg the experiment drug or placeble on an empty stomach with 240ml warm water.
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-8 (Sham Comparator): Arm Description: Single ascending-dose study: on day1, subjects will take 800 mg the experiment drug or placeble on an empty stomach with 240ml warm water.
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-9 (Sham Comparator): Multiple ascending-dose study: Day1-Day14 , subjects will take 70 mg, QD experiment drug or placeble with 240ml warm water on an empty stomach.
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-10 (Sham Comparator): Multiple ascending-dose study: Day1-Day14 , subjects will take 150 mg, QD experiment drug or placeble with 240ml warm water on an empty stomach.
  Interventions: Drug: HEC169584 capsule; Drug: placebo
- Dose group-11 (Sham Comparator): Multiple ascending-dose study: Day1-Day14 , subjects will take 300 mg, QD experiment drug or placeble with 240ml warm water on an empty stomach.
  Interventions: Drug: HEC169584 capsule; Drug: placebo

INTERVENTIONS:
Drug: HEC169584 capsule — Each dose of HEC83518 will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
Drug: placebo — The placebo will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  Arms: Dose group-10; Dose group-11; Dose group-2; Dose group-3; Dose group-4; Dose group-5; Dose group-6; Dose group-7; Dose group-8; Dose group-9

SUMMARY:
The safety, tolerability, and pharmacokinetic/pharmacodynamic (PK/PD) characteristics study of HEC169584 capsules in healthy subjects .

DETAILED DESCRIPTION:
This trial adopts a single - center, randomized, double - blind, placebo - controlled, dose - escalation trial design.

This trial is divided into two parts. The first part consists of a single - ascending - dose (SAD) trial and a food - effect (FE) trial. The second part is a multiple - ascending - dose (MAD) tria.

Screening will be conducted within 28 days prior to the first drug administration. After all test results are obtained, inclusion and exclusion criteria will be verified. Eligible subjects will be admitted to the research center one day before drug administration (D - 1). Researchers will assign random numbers to eligible subjects of the same dose group in ascending order according to their screening numbers, and conduct relevant examinations and collect blood, urine, and fecal samples (if necessary) at the time points specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should understand and abide by the research procedures, volunteer to participate, and sign the informed consent form.
2. When signing the informed consent form, subjects should be between 18 and 45 years old (including the boundary values), and both genders are eligible.
3. Male subjects should weigh ≥ 50.0 kg, and female subjects should weigh ≥ 45.0 kg. For the single - dose trial, the body mass index [BMI = weight (kg) / height² (m²)] should be within the range of 18.0 - 28.0 kg/m² (including the boundary values). For the multiple - dose trial, the BMI should be within the range of 18.0 - 30.0 kg/m² (including the boundary values).
4. Subjects enrolled in the MAD (Multiple - Ascending - Dose) trial should also meet the requirement that 2.6 mmol/L (100 mg/dL) ≤ LDL - C < 4.1 mmol/L (160 mg/dL).
5. The results of vital signs, physical examinations, clinical laboratory tests, electrocardiograms, chest X - rays (posteroanterior view), abdominal color Doppler ultrasounds, etc. should be normal, or if judged as abnormal by the investigator, they should be of no clinical significance.
6. Subjects (including their partners) should voluntarily adopt effective contraceptive measures from the screening stage until 3 months after the last drug administration, and should have no plans for sperm or egg donation.

Exclusion Criteria:

1. Subjects had clinically significant diseases as follows (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, neoplastic, pulmonary, immunological, mental, or cardiovascular and cerebrovascular diseases) before screening.
2. Subjects with allergic constitution (allergic to multiple drugs or foods).
3. Subjects who smoked more than 5 cigarettes per day on average within 3 months before screening, or smoked within 48 hours before taking the investigational product, or could not stop using any tobacco products during the trial.
4. Subjects had a history of dysphagia before screening, or had a history of gastrointestinal, hepatic, or renal diseases or surgeries that potentially affect the absorption, distribution, metabolism, and excretion of the investigational product (except uncomplicated appendectomy and hernia repair).
5. Subjects had a history of alcoholism within 1 year before screening (consuming 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine), or had a positive alcohol breath test during the screening period.
6. Subjects had a history of drug abuse or used drugs within 2 years before screening, or had a positive urine drug screening during the screening period.
7. Subjects donated blood or lost blood ≥ 400 mL within 3 months before screening, or planned to donate blood within 1 month after the end of the trial.
8. Subjects had a history of thyroid diseases, or the thyroid - stimulating hormone (TSH) index in the thyroid function test during the screening period was beyond the normal range.
9. Subjects had a corrected QT interval (QTcF = QT/RR0.33 calculated by the Fridericia formula) of the 12 - lead electrocardiogram > 450 ms during screening.
10. Subjects had a glomerular filtration rate < 90 mL/min (the glomerular filtration rate is calculated using the simplified MDRD formula: for men, eGFR = 186 × creatinine (mg/dL)-1.154 × age - 0.203; for women, eGFR = 186 × creatinine (mg/dL)-1.154 × age - 0.203 × 0.742). Note: The unit of creatinine in the formula is mg/dL. When calculating, the creatinine result in μmol/L needs to be converted to mg/dL, and 1 μmol/L = 0.01131 mg/dL.
11. Subjects received vaccination within 1 month before screening, or planned to receive vaccination during the trial.
12. Subjects took inhibitors and/or inducers of CYP3A4, CYP2C8, P - gp, or BCRP within 4 weeks before screening.
13. Subjects took any prescription drugs, over - the - counter drugs, any vitamin products, or Chinese herbal medicines within 14 days before screening.
14. Subjects consumed foods or beverages containing chocolate, caffeine, xanthine, alcohol, or grapefruit within 48 hours before the first drug administration.
15. Subjects developed an acute illness or had concomitant medications from the screening stage to before the first drug administration.
16. Subjects had a history of fainting at the sight of needles or blood, could not tolerate intravenous puncture for blood collection, or had difficulty in blood collection.
17. Lactating or pregnant women, or women of child - bearing potential with a positive pregnancy test.
18. Subjects participated in other clinical trials within 3 months before screening (if the subject withdrew from the study before treatment, that is, was not randomized or did not receive treatment, they can be enrolled in this study).
19. Subjects tested positive for any one of hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, or treponema pallidum antibody.
20. Subjects had special dietary requirements and could not accept the unified diet.
21. Subjects with other factors that, in the investigator's opinion, make them inappropriate to participate in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-08-14 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-06 (Estimated)

PRIMARY OUTCOMES:
Adverse event | up to 27 days
  Evaluate the safety and tolerability of single/multiple administrations of HEC169584 capsules in healthy subjects.

SECONDARY OUTCOMES:
PK parameters - AUC0-∞ | up to 48 hours
  area under the concentration versus time curve (AUC) from time zero to infinity
PK parameters - AUC0-t | up to 48 hours
  Area under the concentration versus time curve (AUC) from time zero to 48 h (AUC0-48 )
PK parameters - Cmax | up to 48 hours
  Maximum Plasma Concentration ( Cmax)
PK parameters - tmax | up to 48 hours
  Time to peak(tmax)
PK parameters - t½ | up to 48 hours
  Apparent terminal elimination half-life(t½)
PK parameters -Vz/F | up to 48 hours
  Apparent volume of distribution(Vz/F)
PK parameters -MRT | up to 48 hours
  The Mean Residence Time#(MRT)
PK parameters -CL/F | up to 48 hours
  The Apparent Clearance (CL/F)
PK parameters -The Accumulation Ratio(R) | up to 15 days
  The Accumulation Ratio(R)
PK parameters -Food Effect on the Cmax | up to 48 hours
  The geometric mean percentage of Cmax between post - meal administration and fasting administration
PK parameters -Food Effect on the AUC | up to 48 hours
  The geometric mean percentage of AUC between post - meal administration and fasting administration
The pharmacodynamics of HEC169584 capsules | Time Frame: up to 28 days
  The pharmacodynamics of HEC169584 capsules was preliminarily explored through SHBG(Sex Hormone - Binding Globulin) and Fasting blood lipid.

OTHER OUTCOMES:
C-QT study, drug metabolism and excretion, drug - drug interaction characteristics (if necessary), pharmacogenomic characteristics (if necessary) | up to 28 days
  Explore the impact of the blood concentration of HEC169584 capsules on the QTc interval.
  Explore characteristics such as drug metabolism and excretion, drug - drug interactions (if necessary), and pharmacogenomic characteristic (if necessary).

CONTACTS AND LOCATIONS:
Overall Officials: DongYang Liu, doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- No. 49, Huayuan North Road, Haidian District, Beijing Municipality, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No